CLINICAL TRIAL: NCT00124462
Title: A Randomized Trial of Realignment Therapy for Treatment of Medial Knee Osteoarthritis
Brief Title: Trial of Realignment Therapy for Treatment of Medial Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: H-24147; H133G040201 (Other Grant/Funding Number: NIDRR)
Record Dates: First submitted 2005-07-26; First posted 2005-07-28 (Estimated); Results first posted 2017-06-29 (Actual); Last update posted 2017-06-29 (Actual); Status verified 2017-05

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Realignment to Placebo (Other): Realigning knee brace and custom orthodic- A valgus brace, customized functional orthotic for neutral foot position and motion control footwear.
  Interventions: Device: Realigning knee brace and custom orthodic; Device: Non realigning knee brace and flat orthodic
- Placebo to Realignment (Other): Non realigning knee brace and flat orthodic- A neutral brace that does not have any varus/valgus angulation, control foot orthodic and shoes with flexible midsole
  Interventions: Device: Realigning knee brace and custom orthodic; Device: Non realigning knee brace and flat orthodic

INTERVENTIONS:
Device: Realigning knee brace and custom orthodic — A valgus brace, customized functional orthotic for neutral foot position and motion control footwear
Device: Non realigning knee brace and flat orthodic — A neutral brace that does not have any varus/valgus angulation, control foot orthodic and shoes with flexible midsole

SUMMARY:
The overall objective of this 3-year project is to determine whether the provision of realignment therapy in patients with medial knee osteoarthritis (OA) relieves knee pain and improves function. The researchers will test the hypothesis that compared to control treatment, the use of realignment therapy (valgus knee brace + motion control shoes + orthosis) is effective in medial knee OA.

The specific aims are:

* To undertake a 30 week randomized crossover clinical trial in patients with medial knee osteoarthritis to determine whether provision of realignment therapy leads to lower pain scores and improved function during the time of this treatment than during the use of a placebo treatment;
* To perform an open label follow-up study to track use and effectiveness of treatment. This project will be co-funded by DonJoy Orthopedic, a knee bracing company.

DETAILED DESCRIPTION:
We propose a double blind, randomized crossover trial of a realignment therapy for patients with medial knee osteoarthritis with the primary outcome being knee pain and function as assessed by the WOMAC Osteoarthritis Index (VAS Version). Because of the possibility that the therapy may provide proprioceptive input and improve symptoms on that basis, we will test two different treatments: 1. CONTROL TREATMENT A) a neutral brace that does not have any varus/valgus angulation, control foot orthotic and shoes with flexible midsole and 2. ACTIVE TREATMENT B) an valgus brace, customized functional orthotic for neutral foot position and motion control footwear. A run-in design will be used to maximize the likelihood of recruiting subjects who will remain in the trial. Subjects will be randomized to treatment A or B for 12 weeks. We will then remove the realignment therapy of treatment period 1, and they will have no realignment therapy for 6 weeks, after which they will receive the other treatment. For each subject, the trial will last 34 weeks. Study evaluation will take place at the Boston University Medical Center GCRC. The trial will be followed by a 6-month open-label follow up. Trial Schedule. We plan a study lasting a total of 30 weeks from the time of randomization for all subjects. There will be 4 weeks pre-randomization for run-in; a phone call at -4weeks and a visit at -2 weeks. The schedule of visits is shown in the protocol as is the timeline. Intervention The active treatment brace will be the DonJoy OA valgus brace. The active treatment orthosis will consist of a customized functional orthosis to achieve neutral foot position. The active treatment shoewear will be a motion control shoe with an appropriate (based upon foot posture examination) density midsole and heel counter. The control treatment brace will consist of an identical brace with a loosened screw at the hinge allowing varus-valgus laxity. The control treatment orthosis will be flat 1/8" thick inserts of an identical material to the active treatment arm. The control treatment shoe will be identical in appearance with a low density midsole to limit motion control. Treatment shoes will be worn on both feet during each treatment period. Recruitment One key element ensuring success in recruitment for the proposed clinical trial for osteoarthritis is experience with and history of success in recruitment for previous studies. We have successfully recruited targeted number of subjects for 2 recent OA clinical trials and a natural history study of OA all of which have more subjects than are targeted here. We are currently completing an NIH-funded heel wedge study which uses a similar design and study population to the one being employed here and both the clinical trial experience obtained, and the continuing recruitment for that study will facilitate recruitment for this trial. The efficacy of a clinical trial is maximized if subjects comply with assigned treatment and come to scheduled visits. One way to increase the likelihood of subject compliance with a trial is to perform a run-in test, a period of observation prior to randomization during which subjects get experience with major components of the study protocol. Those subjects who have trouble complying with the protocol are excluded before being randomized. Despite the exclusion of potential subjects, trial run-ins have been shown to enhance a trial's statistical power by limiting its results to those who were especially likely to actually receive treatment. A recent test of a run-in in an osteoarthritis trial reported that roughly 10% failed a 4-week run-in and that the exclusion of these subjects from the trial increased efficiency and lowered the number of subjects needed and was highly beneficial. We propose a run in period in which there will be a screening phone call, a visit two weeks later (prerandomization visit), with the randomization visit 2 weeks after the initial visit. This will be a placebo run-in with administration of the control shoe and orthotic for this 2-week period. The run in serves several purposes in addition to the efficiency and adherence reasons noted above. It permits us to obtain radiographs, assess and custom manufacture knee brace, orthotics and shoewear, and review them prior to randomization. It also allows us to assess pain status twice so as to get an average of knee pain scores prior to the trial. One concern of a run-in is that it may limit generalizability by excluding some subjects who fail the run-in test. In this trial we will be assessing efficacy so we need to maximize internal validity. Moreover losing subjects in crossover trial is a major concern and we would like to minimize this. We will preserve allocation concealment by having the randomization codes held by the Data Coordinating Center at Boston University, School of Public Health that is external to the Clinical Epidemiology and Research Training Unit. We will stratify patients into those with end stage (Kellgren & Lawrence Grade 4-specifically bone on bone in the weight bearing knee film in the medial compartment) versus those with disease that is moderate or mild yet still affecting the medial joint. We will then perform blocked stratified randomization ensuring that we randomize roughly equal numbers of patients with severe disease and those with mild to moderate diseases into each of the two treatment arms. We will incorporate a blocked randomization scheme so as to permit roughly equal numbers of subjects to be randomized to each treatment within each of the strata of interest. Blinding We will attempt to conduct a blinded trial. Ideally, a blinded trial presents identical appearing treatments to the patients, and obviously, we cannot accomplish this. Nonetheless, our description of the treatments to the patients will be that we will be comparing two types of treatment for their knee arthritis without specifying which therapy constitutes active treatment. The physician responsible for observations during the study visits will also be blind to subject interventions during each phase. Outcomes to be assessed -Primary Outcome -WOMAC Pain and Function Subscales (Most symptomatic treated Knee) -Secondary Outcomes WOMAC Stiffness Subscale Knee Injury and Osteoarthritis Outcome Score Patient Global Assessment Overall Knee Pain V.A.S. (Knee specific) SF36 Analgesic Use (Medication log) Blinded knee exam by physician Physician Global Assessment Functional performance measures (timed gait and chair stand) Gait analysis (see further description below) Knee malalignment (Measured from long limb films) Proprioception (Ability to reproduce passive positioning of the knee). Open Label Follow-up At the end of their participation in the trial, subjects will be allowed to keep the therapy they used. We will ask them which therapy helped them most, and we will strongly encourage continued use. We will continue to follow these subjects for an additional 6 months. We will schedule open label study follow-up visits at 2, 4 and 6 months during which subjects' realignment therapy will be re-examined. Replacements will be provided if necessary. We will also administer the WOMAC at these visits to asses whether treatment effects remain. At these visits, subjects will be queried about adherence; whether they continue to use the realignment therapy, how many days per week (from an adherence diary) they have worn them. This data will enable an assessment of long term adherence, and also enable us to ascertain if response is contingent on adherence. During all phases of the study participation, subjects will receive educational materials that have been approved by the IRB either during their visits or via the mail. These are intended to keep subjects engaged and thereby help with retention in the study.

ELIGIBILITY:
Inclusion Criteria:

* Trial participants must meet American College of Rheumatology (ACR) criteria for osteoarthritis with knee pain, aching or stiffness on most of the past 30 days and evidence on radiograph of a definite osteophyte. In addition, because the researchers are interested in recruiting persons with medial knee osteoarthritis, participants will need to have evidence of disease in this compartment on their radiographs, and not have lateral compartment or patellofemoral compartment disease. Medial disease is based on definitions used in the researcher's previous publications as definite radiographic OA + at least grade 1 medial narrowing (0-3 scale) using an atlas from the Osteoarthritis Research Society International.

Exclusion Criteria:

* Individuals with clinical evidence of patellofemoral disease or knee pathology (other than medial compartment OA) likely to be causing their knee pain.
* Individuals who usually use an ambulation aid to walk such as a cane, crutch, walker or wheel chair.
* Amputation of foot or previous major trauma to foot that would raise concerns about whether an insert might worsen foot pain. Persons with foot lesions such as sores or ulcers in which redistributing load in the foot might be dangerous, will be excluded.
* Known neuropathy from diabetes or for other reasons.
* Past history of deep venous thrombosis.
* Pain emanating more from back or hip than from knee as determined by screening questionnaire
* Low pain score on WOMAC, a widely used and well validated questionnaire to assess knee symptoms. To evaluate response, the researchers will require that patients have a minimal score of at least 4 out of 10 on at least 2 of 5 questions, or a total of greater than 15 out of 50 for the WOMAC pain scale in the eligible knee at pre-randomization phone call and visit, and at randomization visit. This will allow us to detect response to treatment if response occurs.
* Planning to move from area within 9 months of study screening
* Symptomatic comorbid disease limits walking more than knee pain (per screening questionnaire)
* Receiving corticosteroid injections in the month prior to starting the trial. No other treatments will trigger exclusion, although for patients who have been on glucosamine +/or chondroitin +/or nonsteroidal anti-inflammatory drug (NSAID) the researchers will require that they must have taken these treatments for at least 2 months prior to onset of trial and to commit to not start a new treatment throughout the trial.
* Bilateral total knee replacements (TKR) or plan for TKR in next 6 months for affected knee.
* Known other causes of arthritis including rheumatoid arthritis (RA), systemic lupus erythematosus (SLE), gout, psoriatic arthritis, pseudogout.
* Failure to pass 4 week run-in test.
* Volunteers in a pre-contemplative state (persons who would not consider realignment therapy as a therapeutic option for their knee OA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2008-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Hunter, Principal Investigator — Boston University
Locations (1):
- Boston University, School of Medicine, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects will be recruited from: 1) various different forms of public media including Boston Globe, Baystate Banner. 2) BMC patients referred from colleagues in the rheumatology and orthopedic sections. 3) individuals already recruited for other clinical trials with consent forms that included permission to call subjects for other studies)
Groups:
- Realignment to Placebo: Realignment/Experimental Knee Brace and Shoe Insert- A valgus brace, customized functional orthodic for neutral foot position and motion control footwear.
  Placebo/Control Knee brace and Shoe Insert- A neutral brace that does not have any varus/valgus angulation, control foot orthodic and shoes with flexible midsole
- Placebo to Realignment: Placebo/Control Knee brace and Shoe Insert- A neutral brace that does not have any varus/valgus angulation, control foot orthodic and shoes with flexible midsole.
  Realignment/Experimental Knee Brace and Shoe Insert- A valgus brace, customized functional orthodic for neutral foot position and motion control footwear.
Period: Overall Study
Arm/Group | Realignment to Placebo | Placebo to Realignment
Started | 40 | 40
Completed | 29 | 27
Not Completed | 11 | 13
Not completed — Lost to Follow-up | 3 | 3
Not completed — Physician Decision | 3 | 4
Not completed — Withdrawal by Subject | 4 | 5
Not completed — Device fitting, n=2, other hlth issues | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Realignment to Placebo: Realigning knee brace and custom orthodic: A valgus brace, customized functional orthotic for neutral foot position and motion control footwear Non realigning knee brace and flat orthodic: A neutral brace that does not have any varus/valgus angulation, control foot orthodic and shoes with flexible midsole
- Total: Total of all reporting groups
Arm/Group | Realignment to Placebo | Placebo to Realignment | Total
Number analyzed (Participants) | 40 | 40 | 80
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (10.8) | 60 (13.1) | 62 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 25 | 50
  Male | 15 | 15 | 30
BMI [Mean (Standard Deviation); unit: kg/m2] — Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. A BMI below 18.5 is underweight, between 18.5 and 24.9 is considered normal weight, 25 to 29.9 is overweight, a BMI 30-34.9 is moderately obese is, and a BMI 35 or greater is obese.
  kg/m2 | 32.7 (8.4) | 34.7 (10.8) | 33.6 (9.4)
WOMAC pain score [Mean (Standard Deviation); unit: units on a scale] — The WOMAC (Western Ontario and McMaster Osteoarthritis Index) is a widely used self-administered health status measure used in assessing pain, stiffness, and function in patients with OA of the hip or knee. It measures Pain (5 questions), Stiffness (2 questions), and Function (17 questions). The WOMAC pain scale ranges from 0-20. All the items are scored on a scale of 0-4 (0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely). Lower scores indicate lower levels of pain.
  units on a scale | 9.2 (3.4) | 9.1 (3.4) | 9.15 (3.4)
WOMAC function score [Mean (Standard Deviation); unit: units on a scale] — The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a self-administered health status measure for pain, stiffness, and function in patients with knee or hip OA. It measures Pain (5 questions), Stiffness (2 questions), and Function (17 questions). The WOMAC function score ranges from 0-68, all items are scored on a scale of 0-4 (0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely) for difficulty of specific functions. Lower overall function scores indicate higher levels of functioning or less difficulty performing a list of 17 specific activities.
  units on a scale | 33.3 (11.8) | 34.6 (10.3) | 33.9 (11.1)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change WOMAC Pain Scale (Most Symptomatic Treated Knee)
Description: The WOMAC (Western Ontario and McMaster Osteoarthritis Index) is a widely used self-administered health status measure used in assessing pain, stiffness, and function in patients with OA of the hip or knee. It measures Pain (5 questions), Stiffness (2 questions), and Function (17 questions). The WOMAC pain scale ranges from 0-20. All the items are scored on a scale of 0-4 (0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely). Lower scores indicate lower levels of pain.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale change from baseline
Arm/Group | Realignment to Placebo | Placebo to Realignment
Number analyzed (Participants) | 29 | 27
units on a scale change from baseline | -2.2 (3.3) | -1.7 (3.8)

2. Primary Outcome: Change in WOMAC Function Scale (Most Symptomatic Treated Knee)
Description: The WOMAC (Western Ontario and McMaster Universities Osteoarthritis Index) is a self-administered health status measure for pain, stiffness, and function in patients with knee or hip OA. It measures Pain (5 questions), Stiffness (2 questions), and Function (17 questions). The WOMAC function score ranges from 0-68, all items are scored on a scale of 0-4 (0 = None, 1 = Slight, 2 = Moderate, 3 = Very, 4 = Extremely) for difficulty of specific functions. Lower overall function scores indicate higher levels of functioning or less difficulty performing a list of 17 specific activities.
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale change from baseline
Arm/Group | Realignment to Placebo | Placebo to Realignment
Number analyzed (Participants) | 29 | 27
units on a scale change from baseline | -5.1 (12.1) | -4.6 (9.6)

ADVERSE EVENTS:
Groups:
- Placebo to Realignment: Non realigning knee brace and flat orthodic- A neutral brace that does not have any varus/valgus angulation, control foot orthodic and shoes with flexible midsole Realigning knee brace and custom orthodic: A valgus brace, customized functional orthotic for neutral foot position and motion control footwear
Arm/Group | Realignment to Placebo | Placebo to Realignment
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/27
Other Adverse Events (participants affected / at risk) | 0/29 | 0/27

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes